CLINICAL TRIAL: NCT01298323
Title: A Randomized,Int.,Open-Label Phase III Study to Assess the Effect of a Patient Outreach Program on the Percentage of Time Patients With Locally Advanced or Metastatic MTC Experience Grade 2 or Higher AEs in the First 12 Months of Treatment With Vandetanib
Brief Title: Study to Determine if Contacting Patients With MTC More Frequently Results in Earlier Detection and Treatment of Signs and Symptoms of AEs and Thus a Decrease in the Percentage of Time Patients Experience AEs During First 12 Months on Vandetanib Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D4200C00088; LPS14815 (Other: Sanofi Identifier); 2010-023428-26 (EudraCT Number)
Record Dates: First submitted 2011-02-16; First posted 2011-02-17 (Estimated); Results first posted 2014-11-24 (Estimated); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Locally Advanced or Metastatic Medullary Thyroid Cancer; Medullary Thyroid Cancer
Keywords: Medullary Thyroid Cancer; Locally advanced; Metastatic; Vandetanib; Patient Outreach
MeSH Terms: conditions — Carcinoma, Medullary; Neoplasm Metastasis | interventions — vandetanib

ARMS (2):
- Vandetanib Control (Active Comparator): Control - treatment 300mg vandetanib opel label
  Interventions: Drug: Vandetanib
- Experimental (Experimental): Experimental - treatment 300mg vandetanib opel label
  Interventions: Behavioral: Patient outreach; Drug: Vandetanib

INTERVENTIONS:
Behavioral: Patient outreach — Patients will be contacted at week 1 and then every 2 weeks until completion of 52 weeks to detect/treat AEs sooner
  Arms: Experimental
Drug: Vandetanib — Treatment 300mg vandetanib opel label.
  Other Names: SAR390530

SUMMARY:
The purpose of this study is to evaluate the effect of patient outreach program on the proportion of time patients with MTC experience moderate or severe AEs during first 12 months of treatment with vandetanib

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Female or male aged 18 years and over
* Previously confirmed histological diagnosis of unresectable, locally advanced or metastatic hereditary or sporadic MTC. Documentation must be provided in patient's medical chart
* WHO or ECOG Performance status 0-2
* Negative pregnancy test (urine or serum) for female patients of childbearing potential

Exclusion Criteria:

* Unstable brain metastases or spinal cord compression that require treatment, unless treated at least 4 weeks before first dose and stable without steroid treatment for 10 days
* Major surgery within 4 weeks before randomization
* The last dose of prior chemotherapy received less than 3 weeks prior to randomization
* Radiation therapy not completed prior to the first dose of vandetanib
* Significant cardiac event, superior vena cava syndrome, NYHA classification of heart disease ≥2, within 12 weeks before randomization, or presence of cardiac disease that in the opinion of the Investigator increases risk of ventricular arrhythmia
* Creatinine clearance <30 ml/min (calculated by Cockcroft-Gault formula),Patients with moderate renal impairment, defined as creatinine clearance ≥30 to <50 ml/min, must start vandetanib at a reduced dose of 200 mg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2011-02-25 (Actual); Primary Completion 2013-04-26 (Actual); Study Completion 2025-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (66):
- Australia (2):
  - Investigational Site Number : 301, St Leonards, New South Wales
  - Investigational Site Number 301, St Leonards
- Austria (2):
  - Investigational Site Number 401, Vienna
  - Investigational Site Number : 401, Vienna
- Belgium (2):
  - Investigational Site Number : 501, Anderlecht
  - Investigational Site Number 501, Brussels
- Brazil (4):
  - Hospital De Clinicas De Porto Alegre Site Number : 701, Porto Alegre, Rio Grande do Sul
  - Faculdade de Medicina de Ribeirao Preto - USP Site Number : 702, Ribeirão Preto, São Paulo
  - Investigational Site Number 701, Porto Alegre
  - Investigational Site Number 702, Ribeirão Preto
- Bulgaria (2):
  - Investigational Site Number 901, Sofia
  - Investigational Site Number : 901, Sofia
- Canada (6):
  - Investigational Site Number : 1001, London, Ontario
  - Investigational Site Number : 1003, Toronto, Ontario
  - Investigational Site Number : 1002, Sherbrooke, Quebec
  - Investigational Site Number 1001, London
  - Investigational Site Number 1002, Sherbrooke
  - Investigational Site Number 1003, Toronto
- China (4):
  - Investigational Site Number 1301, Beijing
  - Investigational Site Number : 1301, Beijing
  - Investigational Site Number 1302, Shanghai
  - Investigational Site Number : 1302, Shanghai
- Czechia (2):
  - Investigational Site Number 1901, Prague
  - Investigational Site Number : 1901, Prague
- Denmark (2):
  - Investigational Site Number 2001, Odense C
  - Investigational Site Number : 2001, Odense C
- Finland (2):
  - Investigational Site Number 2201, Helsinki
  - Investigational Site Number : 2201, Helsinki
- Germany (6):
  - Investigational Site Number 2602, Essen
  - Investigational Site Number : 2602, Essen
  - Investigational Site Number 2603, Halle
  - Investigational Site Number : 2603, Halle
  - Investigational Site Number 2601, Würzburg
  - Investigational Site Number : 2601, Würzburg
- Greece (2):
  - Investigational Site Number 3001, Athens
  - Investigational Site Number : 3001, Athens
- India (4):
  - Investigational Site Number 3501, Mumbai
  - Investigational Site Number : 3501, Mumbai
  - Investigational Site Number 3502, Vellore
  - Investigational Site Number : 3502, Vellore
- Israel (2):
  - Investigational Site Number 4001, Jerusalem
  - Investigational Site Number : 4001, Jerusalem
- Italy (6):
  - Investigational Site Number 4104, Napoli
  - Investigational Site Number : 4104, Napoli
  - Investigational Site Number 4101, Pisa
  - Investigational Site Number : 4101, Pisa
  - Investigational Site Number 4102, Roma
  - Investigational Site Number : 4102, Roma
- Poland (4):
  - Investigational Site Number : 5702, Poznan, Greater Poland Voivodeship
  - Investigational Site Number : 5703, Warsaw, Masovian Voivodeship
  - Investigational Site Number 5702, Poznan
  - Investigational Site Number 5703, Warsaw
- Russia (6):
  - Investigational Site Number 6201, Moscow
  - Investigational Site Number : 6201, Moscow
  - Investigational Site Number 6204, Moscow
  - Investigational Site Number 6202, Obninsk
  - Investigational Site Number : 6202, Obninsk
  - Investigational Site Number 6203, Saint Petersburg
- South Korea (2):
  - Investigational Site Number : 6001, Seoul
  - Investigational Site Number 6001, Seoul
- Sweden (2):
  - Investigational Site Number 7201, Uppsala
  - Investigational Site Number : 7201, Uppsala
- United Kingdom (4):
  - Investigational Site Number : 2801, Sutton, Surrey
  - Investigational Site Number 2802, Glasgow
  - Investigational Site Number : 2802, Glasgow
  - Investigational Site Number 2801, Sutton

REFERENCES:
- See also: D4200C00088_CSR_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1433&filename=D4200C00088_Study_Synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 25 February 2011 to 27 April 2012, 205 patients were randomized by 33 centers in global 20 countries.
Pre-assignment Details: 217 patients were screened; 205 patients were randomized to treatment.
Groups:
- Vandetanib 300mg; Vandetanib 300mg + Outreach Program: Vandetanib (3 x 100 mg tablet form) was dosed orally, once daily
Period: Overall Study
Arm/Group | Vandetanib 300mg | Vandetanib 300mg + Outreach Program
Started | 102 | 103
Ongoing | 55 | 55
Completed | 16 | 15
Not Completed | 86 | 88
Not completed — Adverse Event | 2 | 4
Not completed — Death | 11 | 16
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Other | 10 | 9
Not completed — Ongoing | 55 | 55
Not completed — Eligibility criteria not fulfilled | 0 | 1

BASELINE CHARACTERISTICS:
Population: Of 103 patients randomized to vandetanib 300 mg+outreach arm, all except 1 patient took part in outreach program . This patient was withdrawn due to eligibility criteria failure and could not be contacted successfully. Hence the results have been summarized under vandetanib 300 mg for safety summaries.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vandetanib 300mg | Vandetanib 300mg + Outreach Program | Total
Number analyzed (Participants) | 102 | 103 | 205
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.8 (13.47) [20 to 77] | 53.0 (14.34) [23 to 77] | 51.9 (13.93) [20 to 77]
Age, Customized [Number; unit: Participants]
  >=18 - <40 Years | 21 | 23 | 44
  >=40 - <65 Years | 65 | 52 | 117
  >=65 - <75 Years | 15 | 22 | 37
  >=75 Years | 1 | 6 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 37 | 75
  Male | 64 | 66 | 130
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 15 | 19 | 34
  White | 87 | 84 | 171

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time a Patient Experienced at Least 1 AE of CTCAE Grade >=2 in First 12 Months of Receiving Vandetanib in Patients Who Participated in Patient Outreach Program.
Description: The primary endpoint is the percentage of time a patient experienced at least one AE of CTCAE grade 2 or higher in the first 12 months of treatment with vandetanib. If the patient discontinues treatment with vandetanib prior to the 12-month time point for any reason, this endpoint will be the time a patient experienced at least one AE of CTCAE grade 2 or higher as a percentage of the time the patient was receiving vandetanib.
Time Frame: 12 months
Population: Number of Months Analyzed is the cumulative sum of number of months that all the participants were present in the study.
Measure: Mean (Standard Deviation); unit: Percentage of days
Units Other Than Participants: months
Groups:
- Vandetanib 300 mg+Outreach Program: Patients on this arm will be contacted by site personnel at week 1 and then every 2 weeks during the first 52 weeks on the study (or prior discontinuation) to detect and possibly treat adverse events sooner than they might have been without the patient outreach, and at a time of lesser CTCAE grade.
- Vandetanib 300 mg: Patients on this arm will get a standard AE monitoring schedule, similar to that used on previous studies. Patients will be asked about any AEs at scheduled visits and will have the option to contact the investigator at any time if experiencing any AE or symptoms and discuss the best treatment options.
Arm/Group | Vandetanib 300 mg+Outreach Program | Vandetanib 300 mg
Number analyzed (Participants) | 102 | 103
Number analyzed (months) | 1513 | 1480
Percentage of days | 51.65 (35.548) [-3.44 to 16.37] | 45.19 (36.347) [-3.44 to 16.37]
Statistical Analysis 1: Comparison: Vandetanib 300 mg+Outreach Program vs Vandetanib 300 mg; Test type: Superiority or Other; p = 0.199, t-test, 2 sided — Statistical significance threshold at this analysis was 10%; t-Statistic = 1.29, 95% CI 2-sided [-3.44 to 16.37]

ADVERSE EVENTS:
Description: Of 103 patients randomized to vandetanib 300 mg+outreach arm, all except 1 patient took part in outreach program . This patient was withdrawn due to eligibility criteria failure and could not be contacted successfully. Hence the results have been summarized under vandetanib 300 mg for safety summaries.
Arm/Group | Vandetanib 300mg | Vandetanib 300mg + Outreach Program
Serious Adverse Events (participants affected / at risk) | 30/103 | 27/102
Other Adverse Events (participants affected / at risk) | 89/103 | 96/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vandetanib 300mg (N=103) | Vandetanib 300mg + Outreach Program (N=102)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Venous insufficiency (Vascular disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Ectopic ACTH syndrome (Endocrine disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 2 (3) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 1 (2) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0)
Death (General disorders) | 2 (2) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis caliciviral (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Haematocrit increased (Investigations) | 1 (1) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Migraine with aura (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Fear (Psychiatric disorders) | 0 (0) | 1 (1)
Azotaemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Glomerulonephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 2 (3)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vandetanib 300mg (N=103) | Vandetanib 300mg + Outreach Program (N=102)
Asthenia (General disorders) | 12 (13) | 12 (14)
Headache (Nervous system disorders) | 8 (9) | 12 (16)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 25 (31) | 26 (28)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 (7) | 4 (4)
Hypothyroidism (Endocrine disorders) | 15 (16) | 15 (16)
Constipation (Gastrointestinal disorders) | 5 (5) | 8 (9)
Diarrhoea (Gastrointestinal disorders) | 48 (63) | 55 (85)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 7 (7)
Nausea (Gastrointestinal disorders) | 19 (21) | 26 (34)
Vomiting (Gastrointestinal disorders) | 11 (13) | 8 (8)
Fatigue (General disorders) | 17 (17) | 18 (19)
Alanine aminotransferase increased (Investigations) | 10 (10) | 9 (9)
Aspartate aminotransferase increased (Investigations) | 8 (8) | 5 (6)
Blood creatinine increased (Investigations) | 8 (9) | 5 (5)
Electrocardiogram QT prolonged (Investigations) | 7 (12) | 9 (13)
Weight decreased (Investigations) | 11 (11) | 12 (12)
Decreased appetite (Metabolism and nutrition disorders) | 19 (20) | 13 (15)
Hypocalcaemia (Metabolism and nutrition disorders) | 14 (18) | 13 (14)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 9 (11)
Dizziness (Nervous system disorders) | 3 (4) | 7 (8)
Dysgeusia (Nervous system disorders) | 6 (6) | 0 (0)
Anxiety (Psychiatric disorders) | 7 (7) | 4 (4)
Insomnia (Psychiatric disorders) | 9 (9) | 8 (10)
Proteinuria (Renal and urinary disorders) | 8 (8) | 11 (15)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6)
Acne (Skin and subcutaneous tissue disorders) | 10 (11) | 7 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (8) | 2 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 22 (23) | 22 (24)
Dry skin (Skin and subcutaneous tissue disorders) | 12 (12) | 7 (8)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 (6) | 5 (5)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 7 (8) | 13 (18)
Hypertension (Vascular disorders) | 31 (35) | 35 (40)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.